CLINICAL TRIAL: NCT04253340
Title: Study of a Bone Assessment Technique, Bone Mineral Analyser, Concerning the Prediction of Improvement in Bone Status After an Infusion of Zoledronic Acid in Osteoporotic Women
Acronym: TEOBASO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Non-functional BMA machine.
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/183/HP
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone mineral analyser (Experimental): Diagnostic Test: Bone mineral analyser
  high resolution digital radiology (200 µm): D0 + M12 Trabecular Bone Score:D0 + M12 DXA scan:D0 + M12
  Interventions: Diagnostic Test: Bone mineral analyser

INTERVENTIONS:
Diagnostic Test: Bone mineral analyser — high resolution digital radiology (200 µm): D0 + M12 Trabecular Bone Score:D0 + M12 DXA scan:D0 + M12

SUMMARY:
* Collection of epidemiological data
* Biological assessment as part of routine care.
* Measurement of the Hurst coefficient at D0
* Measurement of bone density and TBS on D0
* Zoledronic acid infusion the month following inclusion
* phone call at 1 month (observance of zoledronic acid)
* Measurement of bone density, calculation of the Hurst coefficient at M12

ELIGIBILITY:
Inclusion Criteria:

* Women < 85 years old
* Postmenopausal women (amenorrhea for more than 12 months), a confirmation diagnosis should be obtained (amenorrhea for at least 12 months before the inclusion visit).
* Post-menopausal osteoporosis with one or more severe fractures (upper end of the humerus, femur, or tibia; 3 adjacent ribs; lower end of the femur; thoracic or lumbar spine; pelvis), or T score <-3 which justifies setting up a bisphosphonate treatment
* Affiliated to social security

Exclusion Criteria:

* Contraindication to zoledronic acid (allergy to the product, creatinine clearance <35 ml / min, hypocalcemia, open and unhealed lesions of the soft tissues of the mouth)
* Hormone replacement therapy taken in the last 12 months
* Osteoprotective treatment (bisphosphonates, teriparatide, raloxifene, strontium ralenate or denosumab) taken in the last 12 months
* Secondary osteoporosis: hyperthyroidism, hyperparathyroidism, long-term corticosteroid therapy, hypercorticism, hypogonadism, treatment with anti aromatases / LHRH analogues, neoplastic pathology (solid or hemopathy)
* History of bilateral wrist or femur fracture
* Person deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / guardianship or curatorship
* Patient participating in another trial / having participated in another trial within 6 months

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Hurst coefficient | Day 0
  measured by the BMA

SECONDARY OUTCOMES:
Hurst coefficient | Month 12
  measured by the BMA
bone texture parameters | Day 0
  bone texture parameters measured by Trabecular Bone Score
bone texture parameters | Month 12
  bone texture parameters measured by Trabecular Bone Score
Bone mineral density | Day 0
  Bone mineral density measured by DXA scan
Bone mineral density | Month12
  Bone mineral density measured by DXA scan